CLINICAL TRIAL: NCT00755807
Title: Duloxetine in Patients With Central Neuropathic Pain Due to Multiple Sclerosis.
Brief Title: Duloxetine for Multiple Sclerosis Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11666; F1J-US-HMFR (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-11

CONDITIONS: Multiple Sclerosis
Keywords: Central Neuropathic Pain; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine Hydrochloride (HCI)

INTERVENTIONS:
Drug: Duloxetine Hydrochloride (HCI) — Participants received 30 mg duloxetine (po, QD) for 1 week followed by 5 weeks at 60 mg in the acute placebo-controlled period. If the participant completes the double-blind portion of the trial, the participant will be offered the option to participate in the open-label extension period (given 60, 90, or 120 mg QD for 12 weeks).
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine
Drug: Placebo — Participants received placebo oral (po), once daily (QD) for 6 weeks (acute phase). If the participant completes the 6-week double-blind portion of the trial, the participant will be offered the option to participate in the open-label extension period (given 60, 90, or 120 milligrams [mg] QD for 12 weeks).
  Arms: Placebo

SUMMARY:
This study is designed to primarily assess the efficacy and safety of duloxetine 60-120 mg once daily (QD) compared with placebo on the reduction of pain severity in participants with central neuropathic pain due to Multiple Sclerosis.

DETAILED DESCRIPTION:
Study is a multicenter, randomized, double-blind, parallel, placebo-controlled, 20-week trial with 4 study periods. Participants who screen successfully (Study Period I) will be randomized in a 1:1 fashion to duloxetine 60 mg QD or placebo. Starting with Study Period II, participants will be treated in a double-blind manner for 6 weeks. Participants who complete the 6-week, double-blind period will have the opportunity to participate in a 12-week, open-label, flexible-dose portion of the study (Study Period III). Study Period IV is a taper phase designed to reduce the occurrence of discontinuation adverse events. Participants may enter Study Period IV at any time after Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Have central neuropathic pain due to multiple sclerosis (MS) based on the disease diagnostic criteria
* Adult males or females
* Have a score of 4 or greater on the daily 24-hour average pain score
* Females must test negative for pregnancy at study entry
* Complete the daily diaries for at least 70% of the days of the study
* Participants may continue other prescription and nonprescription analgesic pain medications as long as the dose has been stable for 1 month prior to study entry, and they agree to maintain that stable dose throughout the study Disease Diagnostic Criteria:

  * Diagnosis of MS at least 1 year prior to study entry
  * No MS flares or change in disease treatment for the 3 months prior to study entry
  * Daily pain due to MS for a minimum of 3 months prior to study entry

Exclusion Criteria:

* Are currently in a clinical trial of MS disease-modifying therapy
* Have pain that cannot be clearly differentiated from causes other than MS
* Any current or historical diagnosis of mania, bipolar disorder, psychosis, or schizoaffective disorder
* History of substance abuse or dependence
* Are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 Hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lenexa, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roseville, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bismarck, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akron, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melsbroek, Belgium
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenfield Park, Quebec
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine: Participants received 30 milligrams (mg) duloxetine (oral [po], once daily [QD]) for 1 week followed by 5 weeks at 60 mg in the acute placebo-controlled period. If the participant completes the 6-week double-blind portion of the trial, the participant will be offered the option to participate in the open-label extension period (given 60, 90, or 120 mg QD for 12 weeks).
- Placebo: Participants received placebo po, QD for 6 weeks (acute phase). If the participant completes the 6-week double-blind portion of the trial, the participant will be offered the option to participate in the open-label extension period (given 60, 90, or 120 mg QD for 12 weeks).
Period: Acute Phase
Arm/Group | Duloxetine | Placebo
Started | 118 | 121
Completed | 100 | 109
Not Completed | 18 | 12
Not completed — Adverse Event | 16 | 5
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Open-label Extension Phase
Arm/Group | Duloxetine | Placebo
Started | 100 | 109
Completed | 82 | 93
Not Completed | 18 | 16
Not completed — Adverse Event | 7 | 7
Not completed — Protocol Violation | 5 | 2
Not completed — Lack of Efficacy | 3 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 118 | 121 | 239
Age Continuous [Mean (Standard Deviation); unit: years] | 50.77 (9.67) | 52.67 (9.07) | 51.73 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 93 | 179
  Male | 32 | 28 | 60
Race/Ethnicity, Customized [Number; unit: participants]
  African | 9 | 6 | 15
  Caucasian | 109 | 112 | 221
  Hispanic | 0 | 2 | 2
  Native American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 7 | 7 | 14
  Canada | 4 | 7 | 11
  Poland | 20 | 20 | 40
  United States | 87 | 87 | 174
Multiple Sclerosis (MS) Diagnosis Subtype [Number; unit: participants] — National MS Society diagnosis subtypes:
  Primary progressive: initially progressive disease with no plateaus or remissions; or occasional plateau and acute, minor improvements.
  Progressive-relapsing: initial disease progression, but with clear, acute relapses, with or without full recovery from such relapses over time.
  Relapsing-remitting: clearly defined acute attacks with full or partial recovery; no disease progression between attacks.
  Secondary-progressive: initially relapsing-remitting, then progressive at a variable rate, with possible occasional relapse and minor remission.
  participants
    Primary-Progressive | 10 | 16 | 26
    Progressive-Relapsing | 4 | 6 | 10
    Relapsing-Remitting | 81 | 72 | 153
    Secondary-Progressive | 23 | 27 | 50
Duration of MS [Mean (Standard Deviation); unit: years] — How long the participants have had MS.
  years | 11.05 (7.48) | 11.40 (8.49) | 11.23 (7.99)
Duration of central neuropathic pain (CNP) due to MS (n=118, 120) [Mean (Standard Deviation); unit: years] | 6.18 (5.88) | 7.56 (6.69) | 6.88 (6.33)
Weekly 24-Hour Average Pain [Mean (Standard Deviation); unit: units on a scale] — This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the average pain severity over the last 24 hours. Scores are based on daily assessments recorded by participants in their diaries.
  units on a scale | 6.49 (1.41) | 6.31 (1.33) | 6.40 (1.37)
Brief Pain Inventory (BPI) Average Interference (Duloxetine n=116, Placebo n=119) [Mean (Standard Deviation); unit: Units on a scale] — A self-reported scale that measures interference of pain on average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The average Interference scores range from 0 (does not interfere) to 10 (completely interferes).
  Units on a scale | 5.50 (1.98) | 5.24 (2.01) | 5.37 (2.00)
BPI Average Pain (Duloxetine n=116, Placebo n=119) [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 6.09 (1.50) | 5.91 (1.33) | 6.00 (1.42)
Multiple Sclerosis Quality of Life (MS-QOL-54) Overall Quality of Life Subsection [Mean (Standard Deviation); unit: units on a scale] — The MS-QOL-54 is self-reported and consists of 54 questions covering 12 domains: physical function, role limitations due to physical problems, role limitations due to emotional problems, emotional wellbeing, energy, health perceptions, social function, cognitive function, health distress, satisfaction with sexual function, change in health, and overall quality of life. Each domain score is converted into a 0-100 score based on the individual item responses, with higher scores indicating better health status or functioning. Number of participants (n) for duloxetine=116; placebo=119.
  units on a scale | 58.06 (18.61) | 61.78 (18.80) | 59.94 (18.76)
Expanded Disability Status Scale ([EDSS], n=118, 120) [Median (Standard Deviation); unit: units on a scale] — The EDSS is a method of quantifying disability in multiple sclerosis. The EDSS quantifies disability in 8 Functional Systems (pyramidal, cerebellar, brain stem, sensory, bowel and bladder, visual, cerebral, and other) and allows neurologists to assign a functional system score in each. An EDSS of 0.0 is a normal neurological examination. The scores increase in increments of 0.5 starting with 1.0 (no disability, minimal signs in 1 functional system) to 10.0 (death due to MS).
  units on a scale | 4.00 (2.01) | 4.00 (1.78) | 4.00 (1.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly 24-Hour Average Pain Scores at Week 6 (Acute Phase)
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean, with scores ranging from 0 (no pain) to 10 (worst possible pain). Participants should complete electronic diary each day upon awakening. The 11-point Likert scale was used for assessment of 24-hour average pain and evaluated as weekly means. Scores range from 0 (no pain) to 10 (worst possible pain). The Least Squares Mean (LS Mean) Value was adjusted for investigative site and baseline severity.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine: Participants received 30 milligrams (mg) duloxetine (oral [po], once daily [QD]) for 1 week followed by 5 weeks at 60 mg in the acute placebo-controlled period.
- Placebo: Participants received placebo (po, QD) for 6 weeks (acute phase).
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 103 | 115
units on a scale | -1.83 (0.17) | -1.07 (0.16)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Null hypothesis: no difference between duloxetine and placebo on pain severity reduction as measured by weekly mean of the daily 24-hour average pain scores in participants assessed at 6 weeks. Sample size is determined using 2-sided t-test with significance level of 0.05, and 5% of randomized participants without post-baseline data due to very early discontinuation. With 119 participants per arm, study has approximately 80% power to detect an effect size of 0.375 on treatment group difference; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; Mixed model repeated measures (MMRM):Change from Baseline=Baseline+Treatment+Investigator+Week+Treatment*Week+Baseline*Week,participant random effect

2. Secondary Outcome: Change From Baseline in the Weekly 24-Hour Average Pain Scores up to Week 6 (Acute Phase)
Description: This is a nominal outcome reflecting whether or not a clinically-important efficacy outcome (≥30% or ≥50% pain reduction from baseline) was achieved at endpoint. It is based on a comparison between baseline and endpoint scores on an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Used were the weekly mean of the scores of the average pain severity over the last 24 hours. The weekly averages were based on daily assessments recorded by participants in their diaries.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value. Last-observation-carried-forward (LOCF) imputation was implemented for participants with early discontinuation. Baseline-observation-carried-forward (BOCF) imputation was implemented for participants with early discontinuation.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 115 | 119
participants
  ≥30% Reduction (LOCF) | 47 | 32
  ≥50% Reduction (LOCF) | 26 | 19
  ≥30% Reduction (BOCF) | 44 | 29
  ≥50% Reduction (BOCF) | 24 | 16
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.027, Fisher Exact — P-value is for the 30% Reduction (LOCF). P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.246, Fisher Exact — P-value is for 50% Reduction (LOCF). P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.024, Fisher Exact — P-value is for the 30% Reduction (BOCF). P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.165, Fisher Exact — P-value is for 50% Reduction (BOCF). P-values were not adjusted for multiple comparisons; a priori threshold for statistical significance was 0.05

3. Secondary Outcome: Patient Global Impressions of Improvement Scale (PGI-I) at 6 Weeks
Description: A scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). The Least Squares (LS) Mean Value was adjusted for investigative site and baseline severity.
Time Frame: 6 weeks
Population: Number of randomized participants with at least 1 post-baseline value. Last-observation-carried-forward (LOCF) imputation was implemented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 106 | 116
units on a scale | 3.27 (0.11) | 3.48 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.121, ANOVA — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Analysis of Variance (ANOVA) Model: PGI improvement at Endpoint = Treatment + Investigator; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.06 to 0.49] — The mean difference is for placebo - duloxetine

4. Secondary Outcome: Change From Baseline in the Brief Pain Inventory Severity and Interference Scores (BPI-S/BPI-I) at Week 6 (Acute Phase)
Description: Measures pain severity and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst, least, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing pain interference in past 24 hours, such as general activity, mood, normal work, relations with other people, and sleep. Average interference=average of non-missing scores of individual interference items. Least Squares (LS) Mean Value was adjusted for investigative site and baseline severity.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants received placebo (po, QD) for 6 weeks (acute phase). If the participant completes the 6-week double-blind portion of the trial, the participant will be offered the option to participate in the open-label extension period (given 60, 90, or 120 mg QD for 12 weeks).
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 106 | 116
units on a scale
  BPI Severity for Worst Pain | -1.95 (0.21) | -1.29 (0.20)
  BPI Severity for Least Pain | -1.20 (0.18) | -0.72 (0.17)
  BPI Severity for Average Pain | -1.36 (0.19) | -0.84 (0.17)
  BPI Severity for Pain Right Now | -1.91 (0.21) | -1.02 (0.20)
  BPI Interference for General Activity | -1.81 (0.23) | -1.29 (0.22)
  BPI Interference for Mood | -1.91 (0.24) | -1.25 (0.22)
  BPI Interference for Walking Ability | -1.47 (0.25) | -0.91 (0.24)
  BPI Interference for Normal Work | -1.51 (0.24) | -1.18 (0.22)
  BPI Interference for Relations With Others | -1.72 (0.22) | -1.22 (0.20)
  BPI Interference for Sleep | -2.01 (0.22) | -1.59 (0.21)
  BPI Interference for Enjoyment Of Life | -1.82 (0.24) | -1.65 (0.23)
  BPI Mean Interference Score | -1.77 (0.19) | -1.32 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.016, ANCOVA — P-value is for BPI Severity for Worst Pain score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [0.12 to 1.20] — The mean difference is for placebo - duloxetine
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.043, ANCOVA — P-value is for BPI Severity for Least Pain score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.02 to 0.95] — The mean difference is for placebo - duloxetine
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value is for BPI Severity for Average Pain score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.05 to 0.99] — The mean difference is for placebo - duloxetine
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is for BPI Severity for Pain Right Now score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [0.36 to 1.43] — The mean difference is for placebo - duloxetine
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.083, ANCOVA — P-value is for BPI Interference for General Activity score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.07 to 1.11] — The mean difference is for placebo - duloxetine
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.034, ANCOVA — P-value is for BPI Interference for Mood score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [0.05 to 1.27] — The mean difference is for placebo - duloxetine
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.089, ANCOVA — P-value is for BPI Interference for Walking Ability score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.08 to 1.19] — The mean difference is for placebo - duloxetine
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.291, ANCOVA — P-value is for BPI Interference for Normal Work score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.28 to 0.93] — The mean difference is for placebo - duloxetine
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.077, ANCOVA — P-value is for BPI Interference for Relations With Others score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.06 to 1.05] — The mean difference is for placebo - duloxetine
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.148, ANCOVA — P-value is for BPI Interference for Sleep score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.15 to 0.97] — The mean difference is for placebo - duloxetine
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.582, ANCOVA — P-value is for BPI Interference for Enjoyment Of Life score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.45 to 0.79] — The mean difference is for placebo - duloxetine
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.067, ANCOVA — P-value is for BPI Mean Interference score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.03 to 0.94] — The mean difference is for placebo - duloxetine

5. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity Scale (CGI-S) at 6 Weeks (Acute Phase)
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The Least Squares (LS) Mean Value was adjusted for investigative site and baseline severity.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 111 | 114
units on a scale | -0.67 (0.09) | -0.44 (0.08)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.041, ANCOVA — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [0.01 to 0.45] — The mean difference is for placebo - duloxetine

6. Secondary Outcome: Change From Baseline in the Multiple Sclerosis Quality of Life-54 Instrument (MS-QOL-54) at 6 Weeks (Acute Phase)
Description: A 54 question measure covers 12 domains; assesses mental and physical health. Each domain score is converted into a 0-100 score based on individual item responses; higher scores=better health status. The physical health composite score is a weighted average of the physical health scales, such as physical function, health perceptions, and energy. The mental health composite score is a weighted average of the mental health scales, such as overall quality of life, cognitive function, and health distress. The Least Squares (LS) Mean Value was adjusted for investigative site and baseline severity.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 106 | 116
units on a scale
  Physical Health Composite (N=106, 116) | 6.11 (1.15) | 5.12 (1.08)
  Mental Health Composite (N=106, 116) | 5.81 (1.44) | 4.59 (1.35)
  Physical Health (N=106, 116) | 3.35 (1.51) | 2.65 (1.42)
  Health Perceptions (N=106, 116) | 1.41 (1.39) | 1.35 (1.31)
  Energy Subsection Score (N=106, 116) | 6.54 (1.60) | 6.51 (1.50)
  Role Limitation Due to Physical (N=106, 116) | 11.73 (3.17) | 8.60 (2.97)
  Pain (N=106, 116) | 12.42 (1.72) | 8.84 (1.62)
  Sexual Function (N=106, 116) | 1.30 (2.21) | 1.12 (2.09)
  Social Function (N=106, 116) | 5.02 (1.71) | 6.97 (1.61)
  Health Distress (N=106, 116) | 8.96 (1.76) | 9.34 (1.66)
  Overall Quality Of Life (N=106, 116) | 3.66 (1.34) | 5.43 (1.26)
  Emotional Well-being Subsection Score (N=106, 116) | 4.59 (1.37) | 3.99 (1.29)
  Role Limitation Due to Emotional (N=106, 116) | 6.48 (3.55) | 1.58 (3.33)
  Cognitive Function (N=106, 116) | 6.38 (1.45) | 5.57 (1.36)
  Change in Health (N=106, 116) | 8.23 (2.30) | 6.25 (2.16)
  Satisfaction with Sexual Function (N=102, 112) | 2.66 (2.82) | -1.35 (2.68)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.500, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Physical Health Composite Section score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-3.90 to 1.91] — The mean difference is for placebo - duloxetine
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.512, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Mental Health Composite Section score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-4.87 to 2.44] — The mean difference is for placebo - duloxetine
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.720, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Physical Health Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-4.51 to 3.12] — The mean difference is for placebo - duloxetine
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.973, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Health Perceptions Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-3.58 to 3.46] — The mean difference is for placebo - duloxetine
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.991, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Energy Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-4.07 to 4.02] — The mean difference is for placebo - duloxetine
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.441, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Role Limitation Due to Physical Problems Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -3.14, 95% CI 2-sided [-11.14 to 4.87] — The mean difference is for placebo - duloxetine
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.108, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Pain Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -3.58, 95% CI 2-sided [-7.94 to 0.79] — The mean difference is for placebo - duloxetine
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.948, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Sexual Function Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-5.77 to 5.39] — The mean difference is for placebo - duloxetine
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.374, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Social Function Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 1.96, 95% CI 2-sided [-2.37 to 6.28] — The mean difference is for placebo - duloxetine
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.867, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Health Distress Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-4.10 to 4.87] — The mean difference is for placebo - duloxetine
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.306, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Overall Quality Of Life Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [-1.63 to 5.17] — The mean difference is for placebo - duloxetine
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.733, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Emotional Well-being Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-4.08 to 2.88] — The mean difference is for placebo - duloxetine
Statistical Analysis 13: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.283, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Role Limitation Due to Emotional Problems score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -4.90, 95% CI 2-sided [-13.88 to 4.08] — The mean difference is for placebo - duloxetine
Statistical Analysis 14: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.664, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Cognitive Function Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-4.49 to 2.86] — The mean difference is for placebo - duloxetine
Statistical Analysis 15: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.504, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Change in Health Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-7.81 to 3.85] — The mean difference is for placebo - duloxetine
Statistical Analysis 16: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.270, ANCOVA — P-value is for treatment comparison of change from baseline on MSQOL Satisfaction with Sexual Function Subsection score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -4.02, 95% CI 2-sided [-11.18 to 3.14] — The mean difference is for placebo - duloxetine

7. Secondary Outcome: Number of Participants With Suicidal Behaviors, Ideations, and Acts Based on The Columbia Suicide Severity Rating Scale (C-SSRS) at Week 6
Description: C-SSRS scale captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal behaviors, ideations, and acts are provided. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation. Suicidal act: a "yes" answer to actual attempt or completed suicide.
Time Frame: 6 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 118 | 121
participants
  Suicidal Ideation | 3 | 0
  Suicidal Behavior | 1 | 0
  Suicidal Acts | 1 | 0
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.119, Fisher Exact — P-value is for treatment comparison in number of participants with CSSR-S Suicidal Ideation during first 6 weeks of acute treatment. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.494, Fisher Exact — P-value is for treatment comparison in number of participants with CSSR-S Suicidal Behavior during first 6 weeks of acute treatment. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.494, Fisher Exact — P-value is for treatment comparison in number of participants with CSSR-S Suicidal Acts during first 6 weeks of acute treatment. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05

8. Secondary Outcome: Change From Baseline in the Weekly Mean of Night Pain Scores at Week 6 (Acute Phase)
Description: Weekly mean of the night pain severity scores recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). Participants should complete the electronic diary each day upon awakening. The Least Squares (LS) Mean Value was adjusted for investigative site and baseline severity.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 115 | 119
units on a scale | -1.25 (0.12) | -0.74 (0.12)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Mixed model repeated measures model:Change from Baseline=Baseline+Treatment+Investigator+Week+Treatment*Week+Baseline*Week; participant=random effect

9. Secondary Outcome: Change From Baseline in the Beck Depression Inventory II (BDI-II) Question #9 at Week 6 (Acute Phase)
Description: The BDI-II is completed by the participant to rate the severity of depressive symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63 with higher the score indicating more severe depressive symptoms. Question #9 is suicidal thoughts and wishes with a score ranging from 0 to 3.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 105 | 115
units on a scale | -0.04 (0.39) | -0.03 (0.21)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.662, ANCOVA — P-value is for treatment comparison of change from baseline on BDI-II Question #9 score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.04] — The mean difference is for placebo - duloxetine

10. Secondary Outcome: Number of Participants Who Discontinued During the Acute Phase (by Week 6)
Time Frame: Baseline through 6 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 118 | 121
participants
  Discontinued Due to Any Reason | 18 | 12
  Adverse Event (AE) | 16 | 5
  Protocol Violation | 1 | 3
  Subject Decision | 1 | 2
  Lack of Efficacy | 0 | 1
  Physician Decision | 0 | 1
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.244, Fisher Exact — This is the P-value for Discontinuation Due to Any Reason
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.012, Fisher Exact — This is the P-value for Adverse Event (AE)
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.622, Fisher Exact — This is the P-value for Protocol Violation
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — This is the P-value for Subject Decision
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — This is the P-value for Lack of Efficacy
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — This is the P-value for Physician Decision

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Acute Phase
Description: Summary tables of serious adverse events (SAEs) and all other non-serious adverse events are located in the Reported Adverse Event Module.
Time Frame: Baseline through 6 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 118 | 121
participants
  Adverse Events (AEs) - Any Event | 70 | 59
  Serious Adverse Events (SAEs) - Any Event | 4 | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) Resulting in Discontinuation From Baseline During the Acute Phase
Time Frame: Baseline through 6 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 118 | 121
participants
  Any Adverse Event (AE) | 16 | 5
  Dizziness | 3 | 1
  Somnolence | 2 | 0
  Abdominal discomfort | 1 | 0
  Asthenia | 1 | 0
  Back pain | 1 | 0
  Balance disorder | 0 | 1
  Fear | 1 | 0
  Feeling jittery | 1 | 0
  Headache | 0 | 1
  Hypotension | 0 | 1
  Libido decreased | 1 | 0
  Mood altered | 0 | 1
  Nausea | 1 | 0
  Pain in extremity | 1 | 0
  Rash maculo-papular | 1 | 0
  Suicide attempt | 1 | 0
  Throat irritation | 1 | 0

13. Other Pre Specified Outcome: Change From Baseline in Bicarbonate (HCO3) at Week 6 (Acute Phase)
Description: Change from baseline to acute phase endpoint in laboratory assessment for bicarbonate, HCO3.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: milliEq/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 110 | 116
milliEq/Liter
  Baseline | 22.43 (3.01) | 23.23 (2.81)
  Change to Last Observation | 2.08 (2.91) | 1.38 (2.97)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.047, ANOVA — P-value is for treatment comparison of change from baseline on Bicarbonate, HCO3. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Rank-transformed change from Baseline = Treatment + Investigator

14. Other Pre Specified Outcome: Change From Baseline in Creatinine at Week 6 (Acute Phase)
Description: Change from baseline to acute phase endpoint in laboratory assessment of creatinine.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 116
milligram/deciliter (mg/dL)
  Baseline | 0.79 (0.15) | 0.78 (0.17)
  Change to Last Observation | -0.00 (0.20) | 0.01 (0.09)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.033, ANOVA — P-value is for treatment comparison of change from baseline on creatinine. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Rank-transformed change from Baseline = Treatment + Investigator

15. Other Pre Specified Outcome: Change From Baseline in the Platelet Count at Week 6 (Acute Phase)
Description: Change from baseline to acute phase endpoint in laboratory assessment of platelet count.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: Thousand/microliter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 106 | 113
Thousand/microliter
  Baseline | 266.92 (77.19) | 281.22 (66.78)
  Change to Last Observation | -2.20 (43.10) | -11.00 (40.65)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.034, ANOVA — P-value is for treatment comparison of change from baseline on platelet count. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Rank-transformed change from baseline = Treatment + Investigator

16. Other Pre Specified Outcome: Change From Baseline in Inorganic Phosphorus at Week 6 (Acute Phase)
Description: Change from baseline to acute phase endpoint in laboratory assessment of inorganic phosphorus.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 116
mg/dL
  Baseline | 3.63 (0.60) | 3.68 (0.54)
  Change to Last Observation | -0.17 (0.50) | 0.01 (0.56)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.007, ANOVA — P-value is for treatment comparison of change from baseline on inorganic phosphorus. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Rank-transformed change from Baseline = Treatment + Investigator

17. Other Pre Specified Outcome: Change From Baseline in Uric Acid at Week 6 (Acute Phase)
Description: Change from baseline to acute phase endpoint in laboratory assessment of uric acid.
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 110 | 116
mg/dL
  Baseline | 5.19 (1.58) | 4.74 (1.30)
  Change to Last Observation | -0.23 (0.67) | -0.04 (0.60)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.025, ANOVA — P-value is for treatment comparison of change from baseline on uric acid. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Rank-transformed change from Baseline = Treatment + Investigator

18. Secondary Outcome: Change From Baseline in Blood Pressure at Week 6 (Acute Phase)
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 112 | 119
mm Hg
  Diastolic Blood Pressure | 1.34 (0.66) | 0.48 (0.63)
  Systolic Blood Pressure | 0.34 (1.14) | -0.06 (1.09)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.322, ANCOVA — P-value is for treatment comparison of change from baseline on diastolic blood pressure. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-2.55 to 0.84] — The mean difference is for placebo - duloxetine
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.787, ANCOVA — P-value is for treatment comparison of change from baseline on systolic blood pressure. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-3.32 to 2.52] — The mean difference is for placebo - duloxetine

19. Secondary Outcome: Change From Baseline in Pulse Rate at Week 6 (Acute Phase)
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 112 | 118
beats per minute (bpm) | 1.76 (0.84) | 0.22 (0.81)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.160, ANCOVA — P-value is for treatment comparison of change from baseline on pulse rate. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-3.70 to 0.61] — The mean difference is for placebo - duloxetine

20. Secondary Outcome: Change From Baseline in Weight at Week 6 (Acute Phase)
Time Frame: Baseline, 6 weeks
Population: Number of randomized participants with baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 99 | 115
kilograms (kg) | -0.69 (0.20) | 0.08 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value is for treatment comparison of change from baseline on weight. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Model: Change from Baseline = Treatment + Investigator + Baseline Value; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [0.27 to 1.26] — The mean difference is for placebo - duloxetine

21. Secondary Outcome: Patient Global Impressions of Improvement Scale (PGI-I) Score at 18 Weeks
Description: A scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The scores range from 1 (very much better) to 7 (very much worse).
Time Frame: 18 weeks
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine: All participants randomized to placebo or duloxetine in the acute phase took duloxetine during extension phase: 60, 90, or 120 mg QD for 12 weeks (open-label extension phase).
Arm/Group | Duloxetine
Number analyzed (Participants) | 204
units on a scale | 2.67 (1.25)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean PGI-I score at 18 weeks for all participants who entered extension phase

22. Secondary Outcome: Change From Baseline in Brief Pain Inventory Severity and Interference Scores (BPI-S/BPI-I) at Week 18
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
Time Frame: Baseline (end of acute phase/Week 6), Endpoint (Week 18)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 201
units on a scale
  BPI-S for Worst Pain | -1.27 (2.07)
  BPI-S for Least Pain | -0.96 (1.84)
  BPI-S for Average Pain | -1.26 (1.76)
  BPI-S for Pain Right Now | -1.03 (2.20)
  BPI-I for General Activity | -1.01 (2.50)
  BPI-I for Mood | -1.08 (2.56)
  BPI-I for Walking Ability | -0.84 (2.62)
  BPI-I for Normal Work | -1.00 (2.60)
  BPI-I for Relations With Others | -0.65 (2.59)
  BPI-I for Sleep | -0.70 (2.37)
  BPI-I for Enjoyment Of Life | -1.03 (2.47)
  BPI for Mean Interference Score | -0.89 (2.06)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for BPI-S for Worst Pain. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-S for Worst Pain
Statistical Analysis 2: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for BPI-S for Least Pain. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-S for Least Pain score
Statistical Analysis 3: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for BPI-S for Average Pain. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-S for Average Pain score
Statistical Analysis 4: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-S for Pain Right Now score
Statistical Analysis 5: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for BPI-I for General Activity. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-I for General Activity score
Statistical Analysis 6: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for the BPI-I for Mood. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-I for Mood score
Statistical Analysis 7: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for the BPI-I for Walking Ability. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-I for Walking Ability score
Statistical Analysis 8: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for the BPI-I for Normal Work. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-I for Normal Work score
Statistical Analysis 9: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for the BPI-I for Relations With Others. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from baseline to endpoint on BPI-I for Relations With Others score
Statistical Analysis 10: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for the BPI-I for Sleep. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-I for Sleep score
Statistical Analysis 11: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for the BPI-I for Enjoyment of Life. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI-I for Enjoyment Of Life score
Statistical Analysis 12: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P-value is for the BPI for Mean Interference Score. P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on BPI for Mean Interference score

23. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity Scale (CGI-S) Score at Week 18 (Open-label Extension Phase)
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 206
units on a scale | -0.59 (1.02)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on CGI-S score for all participants who entered extension phase

24. Secondary Outcome: Change From Baseline in Multiple Sclerosis Quality of Life-54 Instrument (MS-QOL-54) at Week 18 (Open-label Extension Phase)
Description: A 54 question measure covers 12 domains; assesses mental and physical health. Each domain score is converted into a 0-100 score based on individual item responses; higher scores=better health status. The physical health composite score is a weighted average of the physical health scales, such as physical function, health perceptions, and energy. The mental health composite score is a weighted average of the mental health scales, such as overall quality of life, cognitive function, and health distress.
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 201
units on a scale
  Physical Health Composite Section Score (N=198) | 2.70 (12.32)
  Mental Health Composite Section Score (N=201) | 1.97 (14.45)
  Physical Health Subsection Score (N=201) | 3.16 (14.29)
  Health Perceptions Subsection Score (N=201) | 2.24 (14.04)
  Energy Subsection Score (N=201) | 2.93 (15.42)
  Role Limitation Due to Physical Problems (N=201) | 0.50 (39.29)
  Pain Subsection Score (N=201) | 7.45 (17.57)
  Sexual Function Subsection Score (N=198) | 0.79 (23.38)
  Social Function Subsection Score (N=201) | 2.53 (18.30)
  Health Distress Subsection Score (N=201) | 1.44 (18.51)
  Overall Quality Of Life Subsection Score (N=201) | 1.47 (11.04)
  Emotional Well-being Subsection Score (N=201) | 2.63 (13.61)
  Role Limitation Due to Emotional Problems (N=201) | 3.15 (38.96)
  Cognitive Function Subsection Score (N=201) | -0.07 (14.64)
  Change in Health Subsection Score (N=201) | 4.35 (25.30)
  Satisfaction with Sexual Function Subsect (N=195) | 1.92 (30.56)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Physical Health Composite Section score
Statistical Analysis 2: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.054, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Mental Health Composite Section score
Statistical Analysis 3: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Physical Health Subsection score
Statistical Analysis 4: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.025, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Health Perceptions Subsection score
Statistical Analysis 5: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.008, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Energy Subsection score
Statistical Analysis 6: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.858, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Role Limitation Due to Physical Problems Subsection score
Statistical Analysis 7: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Pain Subsection score
Statistical Analysis 8: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.637, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Sexual Function Subsection score
Statistical Analysis 9: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.051, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Social Function Subsection score
Statistical Analysis 10: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.270, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Health Distress Subsection score
Statistical Analysis 11: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.061, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Overall Quality Of Life Subsection score
Statistical Analysis 12: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.007, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Emotional Well-being Subsection score
Statistical Analysis 13: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.253, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Role Limitation Due to Emotional Problems score
Statistical Analysis 14: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.942, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Cognitive Function Subsection score
Statistical Analysis 15: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.016, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Change in Health Subsection score
Statistical Analysis 16: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.381, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on MSQOL Satisfaction with Sexual Function Subsection score

25. Secondary Outcome: Number of Participants With Suicidal Behaviors, Ideations, and Acts Based on The Columbia Suicide Severity Rating Scale (C-SSRS) at Week 18
Description: as for outcome 7
Time Frame: 18 weeks
Population: All randomized participants who entered the extension phase.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 209
participants
  Suicidal Ideation | 1
  Suicidal Behavior | 0
  Suicidal Acts | 0

26. Secondary Outcome: Change in the Weekly Mean of the Night Pain Scores From Week 6 Through Week 18 (Open-label Extension Phase)
Description: Weekly mean of the night pain severity scores recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). Participants should complete the electronic diary each day upon awakening. Each weekly mean change represents change relative to week 6, the baseline of the extension phase.
Time Frame: Baseline (6 weeks) through Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 206
units on a scale
  Week 7 (n=185) | -0.05 (0.07)
  Week 8 (n=205) | -0.31 (0.07)
  Week 9 (n=184) | -0.54 (0.08)
  Week 10 (n=197) | -0.62 (0.08)
  Week 11 (n=166) | -0.75 (0.08)
  Week 12 (n=192) | -0.89 (0.09)
  Week 13 (n=166) | -1.05 (0.09)
  Week 14 (n=177) | -0.98 (0.10)
  Week 15 (n=158) | -0.99 (0.11)
  Week 16 (n=176) | -1.04 (0.11)
  Week 17 (n=156) | -1.11 (0.11)
  Week 18 (n=175) | -1.04 (0.11)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.524, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 7). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Mixed model repeated measures (MMRM) Model: Change from Baseline=Baseline+Investigator+Week+Baseline*Week; participant was treated as random effect
Statistical Analysis 2: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 8). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; MMRM Model: Change from Baseline = Baseline + Investigator + Week + Baseline* Week, where participant was treated as a random effect
Statistical Analysis 3: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 9). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 4: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 10). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 5: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 11). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 6: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 12). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 7: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 13). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 8: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 14). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 9: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 15). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 10: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 16). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 11: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 17). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]
Statistical Analysis 12: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for test of mean change from extension phase baseline to endpoint (Week 18). P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 26, analysis 2]

27. Secondary Outcome: Change From Baseline in Beck Depression Inventory II (BDI-II), Question #9 at Week 18 (Open-label Extension Phase)
Description: The BDI-II is completed by the participant to rate the severity of depressive symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63 with higher the score indicating more severe depressive symptoms. Question #9 is suicidal thoughts and wishes with the score ranging from 0 to 3.
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 200
units on a scale | -0.01 (0.19)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.706, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; 1-sample t-test of mean change from extension phase baseline to endpoint on BDI-II Question #9 score for all participants who entered extension phase

28. Secondary Outcome: Number of Participants Who Discontinued During the Open-label Extension Phase (by Week 18)
Time Frame: Baseline (6 weeks) through Endpoint (18 weeks)
Population: All participants randomized to placebo in acute phase received duloxetine during the extension phase.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 209
participants
  Discontinued Due to Any Reason | 34
  Adverse Event | 14
  Protocol Violation | 7
  Lack of Efficacy | 6
  Subject Decision | 4
  Lost to follow up | 2
  Sponsor Decision | 1

29. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Open-label Extension Phase
Description: as for outcome 11
Time Frame: Baseline (6 weeks) through Endpoint (18 weeks)
Population: All randomized participants in the open-label extension phase.
Measure: Number; unit: participants
Groups:
- Duloxetine: 60 mg oral, once daily (QD) for 6-weeks (acute phase) followed by 60, 90, or 120 mg QD for 12-weeks (open label extension phase).
Arm/Group | Duloxetine
Number analyzed (Participants) | 209
participants
  Adverse Events (AEs) - Any Event | 130
  Serious Adverse Events (SAEs) - Any Event | 7

30. Secondary Outcome: Number of Participants With Adverse Events (AEs) Resulting in Discontinuation During the Open-label Extension Phase
Time Frame: Baseline (6 weeks) through Endpoint (18 weeks)
Population: All randomized participants in the open-label extension phase.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 209
participants
  Due to any AE | 14
  Fatigue | 2
  Somnolence | 2
  Alanine aminotransferase increased | 1
  Constipation | 1
  Diverticulitis | 1
  Dizziness | 1
  Fall | 1
  Hypertension | 1
  Insomnia | 1
  Multiple sclerosis relapse | 1
  Nausea | 1
  Rash pruritic | 1

31. Other Pre Specified Outcome: Change From Baseline in Monocytes at Week 18 (Open-label Extension Phase)
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: Thousand/microliter
Arm/Group | Duloxetine
Number analyzed (Participants) | 198
Thousand/microliter
  Baseline | 0.38 (0.14)
  Change to Last Observation | 0.02 (0.14)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.035, Wilcoxon (Mann-Whitney) — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Wilcoxon signed rank test of mean change from extension phase baseline to endpoint on monocytes

32. Other Pre Specified Outcome: Change From Baseline in Sodium at Week 18 (Open-label Extension Phase)
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: milliEq/Liter
Arm/Group | Duloxetine
Number analyzed (Participants) | 201
milliEq/Liter
  Baseline | 140.08 (3.04)
  Change to Last Observation | -0.36 (2.76)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney) — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Wilcoxon signed rank test of mean change from extension phase baseline to endpoint on sodium

33. Other Pre Specified Outcome: Change From Baseline in Total Protein at Week 18 (Open-label Extension Phase)
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: gram/deciliter (g/dL)
Arm/Group | Duloxetine
Number analyzed (Participants) | 202
gram/deciliter (g/dL)
  Baseline | 7.04 (0.43)
  Change to Last Observation | -0.06 (0.36)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.036, Wilcoxon (Mann-Whitney) — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Wilcoxon signed rank test of mean change from extension phase baseline to endpoint on total protein

34. Secondary Outcome: Change From Baseline in Blood Pressure at Week 18 (Open-label Extension Phase)
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Duloxetine
Number analyzed (Participants) | 207
mm Hg
  Diastolic | -0.58 (8.44)
  Systolic | -1.22 (13.07)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.320, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on diastolic blood pressure
Statistical Analysis 2: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.182, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on systolic blood pressure

35. Secondary Outcome: Change From Baseline in Pulse Rate at Week 18 (Open-label Extension Phase)
Time Frame: Baseline (6 weeks), endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Duloxetine
Number analyzed (Participants) | 207
beats per minute (bpm) | 1.47 (9.81)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.032, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on pulse rate

36. Secondary Outcome: Change From Baseline in Weight at Week 18 (Open-label Extension Phase)
Time Frame: Baseline (6 weeks), Endpoint (18 weeks)
Population: Number of randomized participants who entered and had at least 1 non-missing value during extension phase.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Duloxetine
Number analyzed (Participants) | 190
kilograms (kg) | -0.30 (2.84)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.151, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; One-sample t-test of mean change from extension phase baseline to endpoint on weight

ADVERSE EVENTS:
Groups:
- Duloxetine - Double-Blind Acute Phase: 60 mg oral (po), once daily (QD) for 6 weeks (acute phase)
- Placebo - Double-Blind Acute Phase: Oral, QD for 6 weeks
- Duloxetine - Open-label Extension Phase: Participants previously receiving duloxetine or placebo in the double-blind acute phase received duloxetine 60, 90, or 120 mg QD for 12 weeks (open label extension phase)
Arm/Group | Duloxetine - Double-Blind Acute Phase | Placebo - Double-Blind Acute Phase | Duloxetine - Open-label Extension Phase
Serious Adverse Events (participants affected / at risk) | 4/118 | 0/121 | 7/209
Other Adverse Events (participants affected / at risk) | 70/118 | 59/121 | 130/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine - Double-Blind Acute Phase (N=118) | Placebo - Double-Blind Acute Phase (N=121) | Duloxetine - Open-label Extension Phase (N=209)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine - Double-Blind Acute Phase (N=118) | Placebo - Double-Blind Acute Phase (N=121) | Duloxetine - Open-label Extension Phase (N=209)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (5) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 9 (10) | 7 (7) | 9 (10)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (5)
Fatigue (General disorders) | 9 (9) | 7 (7) | 14 (15)
Feeling jittery (General disorders) | 1 (1) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 5 (6)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 7 (12)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Weight decreased (Investigations) | 4 (4) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 4 (4)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Balance disorder (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 9 (10) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 6 (6) | 7 (7)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 2 (2) | 6 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Somnolence (Nervous system disorders) | 6 (6) | 3 (3) | 6 (6)
Tremor (Nervous system disorders) | 1 (2) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 4 (4)
Libido decreased (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (1)
Thinking abnormal (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days